CLINICAL TRIAL: NCT02681874
Title: Feasibility Study of the Modified-Smart and Secure Children Program in Primary Care
Brief Title: Smart and Secure Children Program for Preschool Obesity
Acronym: SSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of Houston (Other)
Responsible Party: Principal Investigator, Ashley Butler, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-37460; 46486-I (Other Grant/Funding Number: Texas Children's Hospital Pediatric Pilot Award)
Record Dates: First submitted 2016-01-13; First posted 2016-02-15 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: dietary pattern; stress; nutrition; health; obesity; children; minority; pre-schoolers
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Treatment Arm) (Experimental): The Smart and Secure Children (SSC) program is a 10-week manualized intervention that uses a written validated curriculum. The program is group-based and co-led by peer leaders (Parent Leaders). Sessions are 90 minutes. Groups consist of a maximum of five parents. Parent Leaders facilitate conversations on the SSC program content by sharing real life application, experiences, and solutions. Parent Leaders receive a week-long leadership training to deliver the program and will be supervised by the PI who is a licensed clinical psychologist.
  Interventions: Behavioral: SSC Program
- Group B (Control Arm) (Active Comparator): Parents in the control condition will receive the Smart and Secure Children (SSC) program's written handouts. Handouts include didactic curriculum content and instruct parents to write goals and document goal progress.
  Interventions: Behavioral: Written Handouts

INTERVENTIONS:
Behavioral: SSC Program — The Smart and Secure Children (SSC) program is a 10-week manualized intervention that uses a written validated curriculum. The program is group-based and co-led by peer leaders (Parent Leaders). Parent Leaders facilitate conversations on the SSC program content by sharing real life application, experiences, and solutions.
  Arms: Group A (Treatment Arm)
Behavioral: Written Handouts — The handouts are a part of the SSC program that include didactic curriculum content and instruct parents to write goals and document goal progress.
  Arms: Group B (Control Arm)

SUMMARY:
Many behavioral interventions designed to improve dietary patterns for ethnic and racial/minority preschoolers have produced modest outcomes. A limitation of these interventions include a failure to address key factors associated with dietary patterns for these children, such as parental stress levels. Therefore, the identification of intervention models that target these factors and are effective, acceptable, and feasible among parents of young minority children is important.

Subjects will be asked to take part in this study because they are the parents of a child that receives care at a Texas Children's Pediatrics (TCP) clinic where the study is being done and their child's body mass index has been at or above the 85th percentile.

The purpose of this pilot study is to assess the ease and acceptance of providing an intervention for parents of children ages 2-5 years in the pediatric primary care clinic. The purpose is to also assess how well the intervention works in improving the child's dietary patterns.

DETAILED DESCRIPTION:
Thirty (30) subjects will be enrolled across three (3) TCP clinics where the study will take place. Two types of participants will be recruited for this study: parent participants who will receive the intervention and interventionist participants who will deliver the intervention.

Data collected for this study includes 4 types: parent-report questionnaires, parent saliva samples, parent-report of children's 24-hour food recall, and audio-recordings of intervention sessions. Parent-report questionnaires will assess family demographic information, parental stress, depression, and well-being as well as parental feeding practices and child dietary food patterns.

Procedures for Parent Participants:

Parents will be randomized to the intervention (Group A-15 parents) or control condition (Group B-15 parents). Parents who are randomized to the intervention group will then participate in the 10-session SSC program that is co-led by a trained parent interventionist. Sessions will be audio-recorded to allow intervention fidelity checks. Parents who are randomized to the control condition will receive the SSC written handouts, which is enhanced standard of care for parents who are seen in primary care.

If subjects are assigned to Group A, they will participate in ten intervention sessions that are conducted in the TCP clinic. During each session, subjects will be provided with information about specific skills to improve their child's emotional health and dietary patterns and their own stress levels.

If subjects are assigned to Group B, they will receive written handouts about children's dietary patterns and parent stress levels. They will be instructed to write goals and document goal progress. This care plan is the standard practice and is presently implemented in the site's TCP clinics.

After ten weeks, regardless of the group the subjects were assigned to, they will again complete an interview about their child's dietary food patterns and questionnaires about their own emotions/opinions of their parenting and child feeding practices. The subjects will also be asked to collect their saliva at four time points on a single day at home.

Procedures for Interventionist Participants:

Six interventionist participants will be recruited. Those who indicate interest will meet with the PI or a research staff member to obtain consent. They will then receive 40-hours of training in the intervention provided by study staff. Intervention participants will deliver one or more group intervention, which has 10 sessions.

ELIGIBILITY:
Inclusion Criteria for Parent Participants:

* Non-Latino African American or Latino parents/primary caregivers (defined as primary guardian, which may include legal guardians and foster parents) of a child patient (ages 2-5 years) at Texas Children's Pediatrics (TCP) Community Care medical practices (Gulfgate, Cullen, and Corinthian Pointe)
* Parents of children with a body mass index (BMI) of greater than 85th and less than 95th percentile (overweight) and greater than 95th percentile (obese)
* English as the primary household language

Inclusion Criteria for Interventionist Participants:

* Non-Latino African American or Latino, 18 years or older, having a GED/high school diploma, and parent of a young child

Exclusion Criteria for Parent Participants:

* Parents of children with any type of food allergy, parents of children receiving current intervention for weight
* Parents of children with weight-related medical conditions (e.g., Prader-Willi Syndrome)
* Parents of children who are taking medication (e.g.,stimulant) associated with appetite

Exclusion Criteria for Parent Participants:

* None

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2015-12; Primary Completion 2017-12 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Increase in Healthy Food Dietary Patterns | 5 months
  24-hour recalls conducted with parents will be used to assess children's intake of vegetables, fruits, whole grains, and low/non-fat dairy

SECONDARY OUTCOMES:
Decrease in Parental Stress | 5 months
  Parent perceived general stress will be assessed using the Perceived Stress Scale.
Decrease in Parental Stress | 5 months
  Parent perceived parenting stress will be assessed using the Parenting Stress Index-Short Form.
Decrease in Parental Stress | 5 months
  Diurnal cortisol rhythm levels will be determined by obtaining samples of parents' saliva.
Parental Mental Health Improvement | 5 months
  The Center for Epidemiological Depression Studies Scale will be used to determine parental depressive symptoms.
Parental Mental Health Improvement | 5 months
  The Mental Health Continuum-Short Form will be used to measure parents' positive mental health symptoms.
Improvement in Parental Feeding Behaviors | 5 months
  Parental feeding behaviors will be assessed using The Child Feeding Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Butler, Ph.D, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - Texas Children's Pediatric Associates (TCPA), Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Dr. Butler's Profile Page — http://www.texaschildrens.org/find-a-doctor/ashley-michelle-butler-phd